CLINICAL TRIAL: NCT05109039
Title: Effects of Creatine Supplementation on Performance, Body Composition and Mental Health in Female Collegiate Dancers
Brief Title: Creatine Supplementation in Female Collegiate Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Responsible Party: Principal Investigator, Ann Brown, Assistant Professor, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-181
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Creatine
Keywords: creatine, body composition, dancer, cognition
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Supplementation (Experimental)
  Interventions: Dietary Supplement: Creatine
- Placebo Supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine — Participants will consume 0.1g/kg body weight of creatine with 0.1g/kg body weight of maltodextrin for 42 consecutive days
  Arms: Creatine Supplementation
Dietary Supplement: Placebo — Participants will consume 0.2g/kg body weight of maltodextrin for 42 consecutive days
  Arms: Placebo Supplementation

SUMMARY:
This study will be a 6 week creatine supplementation intervention with performance familiarization and pre and post testing. Participants will report to the human performance laboratory (HPL) for baseline to read and sign an informed consent explaining the procedures and potential risks and benefits of participation. Participants will then complete a physical activity readiness questionnaire (PAR-Q) prior to performing any physical tasks. Participants will also be asked to complete testing below in the order described. Participants will become familiar with the pre/post performance tests, which include isokinetic testing, medicine ball throw, vertical jump, and Wingate testing. Twenty-four hours following visit 1, participants will return to the HPL for visit 2 where they will undergo a second familiarization session for the isokinetic testing and Wingate testing only - these two tests require individuals to provide maximal physical efforts and research suggests that participants should perform multiple familiarization trials before beginning experimental trials. At least 72 hours following visit 2, participants will return to the HPL for visit 3 to perform the baseline performance assessments. Following the baseline assessments, participants will be divided into two supplementation groups: creatine and placebo (maltodextrin). These groups will be randomized and matched based on body mass, hours of dance training per week, meat intake, and menstrual cycle phase. Participants will be asked to consume one of the two supplements daily for 42 consecutive days and maintain their regular dance training and eating behaviors. Participants will report to the HPL daily to receive their supplement between the hours of 12pm and 2pm. Following the last day of supplement consumption, participants will report to the HPL to perform post-testing assessments which will be identical to pre testing.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate dance major or minor

Exclusion Criteria:

* Injured within the past 6 months
* Currently consuming creatine supplements

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in fat mass from baseline after 42 days | Change from baseline fat mass at 42 days
  Dual energy x-ray absorptiometry used to assess fat mass (% and kg)
Change in lean mass from baseline after 42 days | Change from baseline lean mass at 42 days
  Dual energy x-ray absorptiometry used to assess lean mass (% and kg)
Change in visceral adipose tissue from baseline after 42 days | Change from baseline visceral adipose tissue at 42 days
  Dual energy x-ray absorptiometry used to assess visceral adipose tissue (cm2)
Change in peak muscular strength from baseline after 42 days | Change from baseline peak muscular strength at 42 days
  Cybex isokinetic dynamometry used to assess peak muscular strength (W)
Change in peak vertical jump height from baseline after 42 days | Change from baseline peak vertical jump height at 42 days
  Cybex isokinetic dynamometry used to assess vertical jump height (in)
Change in upper body muscular power from baseline after 42 days | Change from baseline upper body muscular power at 42 days
  Seated medicine ball toss used to assess upper body muscular power (in)
Change in muscular power from baseline after 42 days | Change from baseline muscular lower at 42 days
  Wingate anaerobic power test used to assess muscular power (W)
Change in depression, anxiety and stress score from baseline after 42 days | Change from baseline depression, anxiety and stress at 42 days
  Depression, anxiety and stress scale (from 0, normal to 42, extremely severe) used to assess depression, anxiety and stress
Change in cognitive performance from baseline after 42 days | Change from baseline cognitive performance at 42 days
  NIH Toolbox for the assessment of Neurological and Behavioral Function ipad application to assess fluid cognitive measures including executive function, attention, episodic memory, processing speed, and working memory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No